CLINICAL TRIAL: NCT01082419
Title: Acoustic Radiation Force Impulse Imaging (ARFI) : a New Technique to Assess Liver Elasticity - Norms in ARFI: Distribution and Reproducibility of ARFI Values in Disease-free Livers or Pathological Livers.
Brief Title: Acoustic Radiation Force Impulse Imaging (ARFI) : a New Technique to Assess Liver Elasticity
Acronym: NARFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2009/21
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Liver Fibrosis; Liver Cirrhosis; Viral Hepatitis; Liver Tumour; Cardiac Failure; Biliary Cholestasis.
Keywords: Liver stiffness measurement; ARFI; fibrosis; hepatopathy
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Heart Failure; Fibrosis; Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group A (Other): healthy volunteers
  Interventions: Device: ARFI measurement
- Group B (Other): patients with supposed disease free liver (normal hepatic and pancreatic biochemistry)
  Interventions: Device: ARFI measurement
- Group D (Other): patients with cirrhosis
  Interventions: Device: ARFI measurement
- Group E (Other): patients with liver tumour and surgery indication
  Interventions: Device: ARFI measurement
- Group F (Other): patients with reversible liver diseases and with acute left cardiac insufficiency
  Interventions: Device: ARFI measurement
- Group C (Other): patients with non cirrhotic hepatopathy
  Interventions: Device: ARFI measurement
- Group G (Other): patients with reversible liver diseases and with biliary cholestasis
  Interventions: Device: ARFI measurement

INTERVENTIONS:
Device: ARFI measurement — ARFI values are measured during a standard liver ultrasound examination, with patient lying on his back and performing a "light" apnea.
  For group A the measurement is made by a second and a third investigator during the same examination.
  Arms: Group A
Device: ARFI measurement — ARFI values are measured during a standard liver ultrasound examination, with patient lying on his back and performing a "light" apnea.
  For all other groups (B, C, D, E) ARFI is measured only once.
  Arms: Group B; Group C; Group D; Group E
Device: ARFI measurement — ARFI values are measured during a standard liver ultrasound examination, with patient lying on his back and performing a "light" apnea.
  For groups F and G : ARFI is measured again after clinical healing.
  Arms: Group F; Group G

SUMMARY:
Liver stiffness measurement (LSM) by non invasive methods is increasingly used to estimate liver fibrosis in patients with chronic liver diseases. However, there is growing evidence that fibrosis is not the only determinant of liver stiffness. Indeed inflammation, cholestasis, congestion could also interfere with stiffness measurements. Acoustic radiation force impulse imaging (ARFI) is a new technology to perform real time LSM. Using a standard ultrasonographic probe, it offers elastography with a flexible metering box at variable depth, allowing the examination of specific area.

DETAILED DESCRIPTION:
There are many causes of chronic liver diseases such as hepatitis C infection, hepatitis B infection, alcohol, NAFLD (non-alcoholic fatty liver disease), drugs and auto-immune liver disease.

Although the causes differ the pathological response to injury tends to be similar leading to fibrosis and cirrhosis.

Liver biopsy is the current gold standard for the assessment of liver fibrosis but is poorly suited for active monitoring because of its expense and morbidity. Thus, development of alternatives that are safe, inexpensive, and reliable is a priority.

Liver stiffness measurement (LSM) by non invasive method is increasingly used to estimate liver fibrosis in patient with chronic liver disease. Acoustic radiation force impulse imaging (ARFI) is a new technology to perform real time LSM. Using a standard ultrasonographic probe, it offers elastography with a flexible metering box at variable depth, allowing the examination of specific area.

The purpose of this work was to evaluate by ARFI, the efficiency of this new technique, the reproducibility inter and intra observer, and the liver elasticity obtained by this method in different patient groups.

The primary endpoint of this work is to evaluate by ARFI, the efficiency of the technique, the reproducibility inter and intra observer, and the elasticity of liver in 6 different patient groups and healthy volunteers.

The different population groups are:

* healthy volunteers Group A
* patients with supposed disease free liver (normal hepatic and pancreatic biochemistry). Group B
* patients with non cirrhotic hepatopathy. Group C
* patients with cirrhosis. Group D
* patients with liver tumour and surgery indication. Group E
* patients with reversible liver diseases:

  * patients with acute left cardiac insufficiency. Group F
  * patients with biliary cholestasis. Group G

ARFI measurements will be performed in a single liver ultrasound exam visit except for patients with reversible liver diseases who will have a second visit with ARFI measurement after clinical healing. The ARFI values are expressed as a speed in m/s.

ELIGIBILITY:
Inclusion Criteria:

* Man or Woman
* Age> 18 years old
* Able to understand the study and to give informed consent
* Informed consent signed by patient and investigator before any study required examination
* With a valid health insurance
* Groups specific inclusion criteria are:
* Group A : healthy volunteers without known liver disease
* Group B : voluntary patients without known liver disease
* Group C and D Patient with a diagnosed chronic liver disease
* Group E : patients with liver tumors (benign or malignant) with surgical indication
* Group F : patients with acute right heart insufficiency diagnosed by a cardiologist
* Group G :patients with biliary cholestasis and imaging evidence of biliary dilatation

Exclusion Criteria:

* Patient under 18 years old
* Not able to understand the study or to give their consent.
* Pregnant woman
* Severe respiratory insufficiency
* Unable to perform a "light" apnea .
* hemodynamic instability (cardiogenic shock, septic or anaphylactic) possibility of disruption of the elasticity and inability to carry patient.
* Chronic heart insufficiency.
* deprived of their liberty by court

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The elasticity parameter will be for each patient the median of ten ARFI values (m/s) in the right liver. | One or two 30 min visit according to the patient group

SECONDARY OUTCOMES:
Inter and intra observer reproducibility | Three 30 min visits in healthy volunteer group.
Median (m/s) of ARFI values between before and after effective treatment for liver reversible disease | From patient admission until patient healing in groups F&G.

CONTACTS AND LOCATIONS:
Overall Officials: Nora FRULIO, Md MSc, Principal Investigator — University Hospital, Bordeaux; Adelaïde Doussau, MD, Msc, Study Chair — University Hospital, Bordeaux
Locations (1):
- University Hospital Bordeaux, Bordeaux, France

REFERENCES:
- [Background] Bonekamp S, Kamel I, Solga S, Clark J. Can imaging modalities diagnose and stage hepatic fibrosis and cirrhosis accurately? J Hepatol. 2009 Jan;50(1):17-35. doi: 10.1016/j.jhep.2008.10.016. Epub 2008 Nov 8. PMID 19022517
- [Background] Castera L, Forns X, Alberti A. Non-invasive evaluation of liver fibrosis using transient elastography. J Hepatol. 2008 May;48(5):835-47. doi: 10.1016/j.jhep.2008.02.008. Epub 2008 Feb 26. PMID 18334275
- [Background] Friedrich-Rust M, Ong MF, Martens S, Sarrazin C, Bojunga J, Zeuzem S, Herrmann E. Performance of transient elastography for the staging of liver fibrosis: a meta-analysis. Gastroenterology. 2008 Apr;134(4):960-74. doi: 10.1053/j.gastro.2008.01.034. Epub 2008 Jan 18. PMID 18395077
- [Background] Ferraioli G, Gulizia R, Filice C. Real-time elastography in the assessment of liver fibrosis. AJR Am J Roentgenol. 2007 Sep;189(3):W170. doi: 10.2214/AJR.07.2318. No abstract available. PMID 17715090
- [Background] Friedrich-Rust M, Ong MF, Herrmann E, Dries V, Samaras P, Zeuzem S, Sarrazin C. Real-time elastography for noninvasive assessment of liver fibrosis in chronic viral hepatitis. AJR Am J Roentgenol. 2007 Mar;188(3):758-64. doi: 10.2214/AJR.06.0322. PMID 17312065